CLINICAL TRIAL: NCT02281058
Title: Open-label Pilot Study of Abatacept for the Treatment of Vitiligo
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Victor Huang, Physician, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014P000699
Record Dates: First submitted 2014-10-29; First posted 2014-11-03 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intervention group (Experimental): Ten subjects recruited to self-administer abatacept 125mg injected subcutaneously weekly for 24 weeks to determine the impact it has on their vitiligo skin lesions.
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — self-injected subcutaneous biologic medication
  Other Names: Orencia

SUMMARY:
Vitiligo is a chronic autoimmune disease with evidence of CTLA-4 involvement. We are performing a pilot study for the treatment of new onset or actively progressing vitiligo with abatacept to determine if weekly self-injections of medication lead to clinical improvement in vitiligo lesions.

DETAILED DESCRIPTION:
Abatacept has been shown to decrease T cell activity and reduce symptoms associated with rheumatoid arthritis. Similar pathways have been shown to be involved in vitiligo. Therefore, we are recruiting 10 adult patients with active vitiligo who meet specific inclusion and exclusion criteria to receive self-administered injections of abatacept weekly starting at week 0 and continuing until week 24. A 32 week follow-up visit will be performed to evaluate secondary endpoints as well. We will be monitoring patients to see if skin lesions of vitiligo stop spreading and start to repigment with continued treatment.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant individuals ages 18 and older with a diagnosis of actively progressive skin lesions of clinically diagnosed vitiligo covering at 5% or great body surface area (defined as development of new lesions or worsening of existing lesions within the past 6 months) not receiving immune suppressive treatment. Both subjects who have received at least one therapy in the past and subjects currently receiving treatment at the time of screening will be eligible providing they undergo a wash out period prior to starting the study (2 weeks for topical agents and systemic agents with short half lives, 1 month for phototherapy)
* Women of childbearing potential (WOCBP) must be using an acceptable method of contraception to avoid pregnancy throughout the study and for up to 10 weeks after the last dose of study drug in such a manner that the risk of pregnancy is minimized
* WOCBP must have a negative serum or urine pregnancy test result (minimum sensitivity 25 IU/L or equivalent units of HCG) within 0 to 48 hours before the first dose of study drug
* Women must not be breast-feeding
* Sexually active fertile men must use effective birth control if their partners are WOCBP

Exclusion Criteria:

* Pregnant or breastfeeding patients
* Patients with segmental, acrofacial, or universal vitiligo
* Patients with evidence of poliosis (white hairs) within the majority (>50%) of their vitiligo lesions
* Patients currently on any other systemic biologic medication, current use of Abatacept, or any other systemic biologic medication within 2 months of study (or within 5 half-lives of last dose of drug)
* Use of systemic immunosuppressive agent within 2 weeks prior to initiation of Abatacept
* Use of potent topical steroids, topical tacrolimus or pimecrolimus within 2 weeks prior to initiation of Abatacept
* Use of phototherapy within one month prior to initiation of Abatacept therapy
* Patients with a history of chronic obstructive pulmonary disease
* History of active Mycobacterium tuberculosis infection (any subspecies) Use of any investigational medication within 28 days prior to enrollment or 5 half-lives if known (whichever is longer)
* Receiving concomitant immune modulating therapy (see concomitant medications, section 8.6). Subjects receiving such agents at screening may be eligible to enroll following a washout period of 2 weeks for topical agents and systemic agents with short half lives
* Subjects who are impaired, incapacitated, or incapable of completing study-related assessments
* Subjects with current symptoms of severe, progressive, or uncontrolled renal, hepatic, hematologic, gastrointestinal, pulmonary, cardiac, neurologic, or cerebral disease, whether or not related to vitiligo and which, in the opinion of the investigator, might place a subject at unacceptable risk for participation in the study
* Subjects with a history of cancer in the last 5 years, other than non-melanoma skin cell cancers cured by local resection or carcinoma in situ. Existing non-melanoma skin cell cancers should be removed, the lesion site healed, and residual cancer ruled out before administration of the study drug
* Subjects who currently abuse drugs or alcohol
* Subjects with evidence (as assessed by the investigator) of active or latent bacterial or viral infections at the time of potential enrollment, including subjects with evidence of human immunodeficiency virus (HIV) detected during screening.
* Subjects with herpes zoster or cytomegalovirus (CMV) that resolved less than 2 months before the informed consent document was signed
* Subjects who have received any live vaccines within 3 months of the anticipated first dose of study medication
* Subjects with any serious bacterial infection within the last 3 months, unless treated and resolved with antibiotics, or any chronic bacterial infection (eg, chronic pyelonephritis, osteomyelitis, or bronchiectasis)
* Subjects at risk for tuberculosis (TB). Specifically excluded from this study will be subjects with a history of active TB within the last 3 years, even if it was treated; a history of active TB greater than 3 years ago, unless there is documentation that the prior anti-TB treatment was appropriate in duration and type; current clinical, radiographic, or laboratory evidence of active TB; and latent TB that was not successfully treated (≥ 4 weeks)
* Subjects must not be positive for hepatitis B surface antigen
* Subjects must not be positive for HIV
* Subjects who are positive for hepatitis C antibody if the presence of hepatitis C virus was also shown with polymerase chain reaction or recombinant immunoblot assay
* Subjects with any of the following laboratory values Hemoglobin < 8.5 g/dL WBC < 3000/mm3 (< 3 x 109/L) Platelets < 100,000/mm3 (< 3 x 109/L) Serum creatinine > 2 times the ULN Serum ALT or AST > 2 times the ULN
* Any other laboratory test results that, in the opinion of the investigator, might place a subject at unacceptable risk for participation in the study
* Allergies to any components of abatacept or its vehicle
* Subjects who have at any time received treatment with any investigational drug within 28 days (or less than 5 terminal half-lives of elimination) of the Day 1 dose
* Any concomitant biologic DMARD, such as anakinra
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-11 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
change in repigmentation with abatacept therapy as measured using the Vitiligo Area and Severity Index (VASI) score | 24 weeks

SECONDARY OUTCOMES:
clinical safety and rate of adverse events as measured by patient-reported side effects | 32 weeks
percentage repigmentation with abatacept therapy as measured using the physician's global assessment | 24 weeks
effect on disease-related quality of life as measured using the validated Vitiligo Quality of Life (VitiQOL) tool | 32 weeks
maintenance of repigmentation after stopping therapy | 32 weeks
initial time to repigmentation | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided